CLINICAL TRIAL: NCT02739594
Title: COMPARE: Comparison of Ibandronate - Zoledronate Regarding Nephrotoxicity in Patients With Multiple Myeloma
Brief Title: Comparison of Ibandronate - Zoledronate Regarding Nephrotoxicity in Multiple Myeloma
Acronym: COMPARE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML18508; 2005-003264-38 (EudraCT Number)
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Results first posted 2016-07-22 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Ibandronic Acid; Zoledronic Acid

ARMS (2):
- Ibandronate (Experimental): Participants with multiple myeloma will be randomized to receive ibandronate every 4 weeks for a planned duration of 92 weeks.
  Interventions: Drug: Ibandronate
- Zoledronate (Active Comparator): Participants with multiple myeloma will be randomized to receive zoledronate every 4 weeks for a planned duration of 92 weeks.
  Interventions: Drug: Zoledronate

INTERVENTIONS:
Drug: Ibandronate — Ibandronate will be administered via 15-minute intravenous (IV) infusion as 6 milligrams (mg) every 4 weeks for 92 weeks.
  Other Names: Bondronat
  Arms: Ibandronate
Drug: Zoledronate — Zoledronate will be administered via 15-minute IV infusion as 4 mg every 4 weeks for 92 weeks.
  Arms: Zoledronate

SUMMARY:
This multicenter, open-label trial will randomize participants with multiple myeloma to a regimen of ibandronate or zoledronate in order to compare the incidence of nephrotoxicity, measured as creatinine clearance (CrCl) reduction greater than (>) 30 percent (%) or an absolute value of 30 milliliters per minute (mL/min) or lower.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed multiple myeloma, Stage II-III as per Salmon and Durie (1975)
* Indication for biphosphonate therapy

Exclusion Criteria:

* Previous therapy with ibandronate or zoledronate within the past 12 months
* Renal insufficiency with serum creatinine >3.0 mg/dL or >265 micromoles per liter (µmol/L) or CrCl <30 mL/min
* Hypersensitivity to ibandronate, zoledronate, or other biphosphonates
* Presence of secondary malignomas, apart from basaliomas and cervical carcinoma in situ
* Severe accompanying illness with organ impairment
* Osteonecrosis of the jaw at the start of the study
* Life expectancy ≤12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2006-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (46):
- Germany (46):
  - Ansbach
  - Aschaffenburg
  - Augsburg
  - Berlin
  - Bremen
  - Cologne
  - Duisburg
  - Erlangen
  - Essen
  - Esslingen am Neckar
  - Frankfurt am Main
  - Göttingen
  - Greifswald
  - Güstrow
  - Gütersloh
  - Halle
  - Hamburg
  - Hamm
  - Hanover
  - Herne
  - Hof
  - Jena
  - Karlsruhe
  - Kassel
  - Koblenz
  - Krefeld
  - Leer
  - Leipzig
  - Ludwigshafen
  - Lübeck
  - Magedburg
  - Minden
  - Moers
  - Mülheim
  - München
  - Münster
  - Neumünster
  - Offenbach
  - Offenburg
  - Oldenburg
  - Stuttgart
  - Tübingen
  - Weiden
  - Wiesbaden
  - Würzburg
  - Zwickau

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibandronate: Participants with multiple myeloma received ibandronate via 15-minute intravenous (IV) infusion as 6 milligrams (mg) every 4 weeks for up to 92 weeks. As a result of slow recruitment, the treatment duration was shortened to 40 weeks for participants who had not yet received 48 weeks of treatment. All participants returned for an additional follow-up observation 4 weeks after the end of treatment.
- Zoledronate: Participants with multiple myeloma received zoledronate via 15-minute IV infusion as 4 mg every 4 weeks for up to 92 weeks. As a result of slow recruitment, the treatment duration was shortened to 40 weeks for participants who had not yet received 48 weeks of treatment. All participants returned for an additional follow-up observation 4 weeks after the end of treatment.
Period: Overall Study
Arm/Group | Ibandronate | Zoledronate
Started | 46 | 43
Completed at Week 44 | 11 | 5
Completed at Week 96 | 10 | 10
Completed | 21 (Includes all participants who reached the protocol-defined end of study (either Week 44 or 96).) | 15 (Includes all participants who reached the protocol-defined end of study (either Week 44 or 96).)
Not Completed | 25 | 28
Not completed — Undesired Event | 3 | 4
Not completed — Violation of Eligibility Criteria | 1 | 2
Not completed — Protocol Violation | 5 | 6
Not completed — Death | 4 | 2
Not completed — Renal Insufficiency | 4 | 6
Not completed — Administrative Reasons | 1 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Elevated Serum Creatinine | 0 | 1
Not completed — Other | 6 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All participants who were randomized and received at least one dose of study medication and for whom at least one measurement of creatinine clearance (CrCl) was obtained.
Groups:
- Ibandronate: Participants with multiple myeloma received ibandronate via 15-minute IV infusion as 6 mg every 4 weeks for up to 92 weeks. As a result of slow recruitment, the treatment duration was shortened to 40 weeks for participants who had not yet received 48 weeks of treatment. All participants returned for an additional follow-up observation 4 weeks after the end of treatment.
- Total: Total of all reporting groups
Arm/Group | Ibandronate | Zoledronate | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (9.4) | 69.1 (9.1) | 67.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Deterioration in Renal Function According to Reduction in Creatinine Clearance (CrCl) From Baseline to Week 44
Description: CrCl was calculated from blood samples using the Cockcroft-Gault formula. Relevant deterioration in renal function was defined as CrCl reduction of 30 percent (%) from Baseline or an absolute value less than or equal to (≤) 30 milliliters per minute (mL/min) at Week 44. The last available value on/before Week 44 was used in the calculation. The percentage of participants with deterioration in renal function at Week 44 was reported.
Time Frame: Baseline, Week 44
Population: Intent-to-Treat (ITT) Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ibandronate | Zoledronate
Number analyzed (Participants) | 41 | 40
percentage of participants | 9.8 [2.7 to 23.1] | 12.5 [4.2 to 26.8]

2. Primary Outcome: Percentage of Participants With Deterioration in Renal Function According to Reduction in CrCl From Baseline to Week 92
Description: CrCl was calculated from blood samples using the Cockcroft-Gault formula. Relevant deterioration in renal function was defined as CrCl reduction of 30% from Baseline or an absolute value ≤30 mL/min at Week 92. The last available value on/before Week 92 was used in the calculation. The percentage of participants with deterioration in renal function at Week 92 was reported.
Time Frame: Baseline, Week 92
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ibandronate | Zoledronate
Number analyzed (Participants) | 41 | 40
percentage of participants | 14.6 [5.6 to 29.2] | 12.5 [4.2 to 26.8]

3. Secondary Outcome: Percentage of Participants With Skeletal-Related Events (SREs)
Description: SREs were defined according to the Bondronat Summary of Product Characteristics (SmPC) to include radiotherapy to bone for treatment of fractures/impending fractures, surgery to bone for treatment of fractures, vertebral fractures, and non-vertebral fractures. The percentage of participants with at least 1 SRE during the study was reported.
Time Frame: From Baseline to end of study (up to Week 96)
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ibandronate | Zoledronate
Number analyzed (Participants) | 41 | 40
percentage of participants | 22.0 [10.6 to 37.6] | 30.0 [16.6 to 46.5]

4. Secondary Outcome: Time to First SRE
Description: SREs were defined according to the Bondronat SmPC to include radiotherapy to bone for treatment of fractures/impending fractures, surgery to bone for treatment of fractures, vertebral fractures, and non-vertebral fractures. Time to first SRE was defined as the time from first dose of study drug to the time of SRE during the study. The median time to first SRE was estimated by Kaplan-Meier analysis and expressed in days.
Time Frame: From Baseline to end of study (up to Week 96)
Population: ITT Population.
Measure: Median (Full Range); unit: days
Arm/Group | Ibandronate | Zoledronate
Number analyzed (Participants) | 41 | 40
days | 393.0 [12 to 727] | 244.5 [21 to 693]

5. Secondary Outcome: Number of SREs for Each Participant
Description: SREs were defined according to the Bondronat SmPC to include radiotherapy to bone for treatment of fractures/impending fractures, surgery to bone for treatment of fractures, vertebral fractures, and non-vertebral fractures. The number of SREs was averaged across all participants, including those participants who did not experience SREs during the study.
Time Frame: From Baseline to end of study (up to Week 96)
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: SREs
Arm/Group | Ibandronate | Zoledronate
Number analyzed (Participants) | 41 | 40
SREs | 0.3 (0.6) | 0.5 (1.1)

6. Secondary Outcome: Percentage of Participants With Osteonecrosis of Jaw
Description: The percentage of participants with at least 1 event of osteonecrosis of jaw during the study was reported.
Time Frame: From Baseline to end of study (up to Week 96)
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ibandronate | Zoledronate
Number analyzed (Participants) | 41 | 40
percentage of participants | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 8.8]

7. Secondary Outcome: Number of Events of Osteonecrosis of Jaw for Each Participant
Description: The number of events of osteonecrosis of jaw was averaged across all participants, including those participants who did not experience the event during the study.
Time Frame: From Baseline to end of study (up to Week 96)
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: events of osteonecrosis of jaw
Arm/Group | Ibandronate | Zoledronate
Number analyzed (Participants) | 41 | 40
events of osteonecrosis of jaw | 0.0 (0.0) | 0.0 (0.0)

8. Secondary Outcome: Percentage of Participants With Zoledronate Dose Reduction
Description: The percentage of participants with at least 1 zoledronate dose reduction during the study was reported.
Time Frame: From Baseline to end of study (up to Week 96)
Population: ITT Population; only the Zoledronate arm was included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zoledronate
Number analyzed (Participants) | 40
percentage of participants | 30.0 [16.6 to 46.5]

9. Secondary Outcome: Number of Zoledronate Dose Reductions for Each Participant
Description: The number of zoledronate dose reductions was averaged across all participants, including those participants who did not have any dose reductions during the study.
Time Frame: From Baseline to end of study (up to Week 96)
Population: ITT Population; only the Zoledronate arm was included.
Measure: Mean (Standard Deviation); unit: dose reductions
Arm/Group | Zoledronate
Number analyzed (Participants) | 40
dose reductions | 0.8 (1.4)

10. Secondary Outcome: Percent Change From Baseline in N-Acetyl-Beta-D-Glucosaminidase (B-NAG)
Description: The percent change in B-NAG was calculated as [Week 44 or 92 B-NAG minus Baseline B-NAG] divided by Baseline B-NAG, multiplied by 100. For the Week 44 analysis, the last available value on/before Week 44 was used in the calculation. For the Week 92 analysis, the last available value on/before Week 92 was used in the calculation.
Time Frame: Baseline and Weeks 44, 92
Population: ITT Population. The "Number of Participants Analyzed" reflects the total number of participants who provided evaluable data for the endpoint.
Measure: Median (Full Range); unit: percent change
Arm/Group | Ibandronate | Zoledronate
Number analyzed (Participants) | 38 | 37
percent change
  Week 44 | -15.7 [-86 to 355] | 10.6 [-94 to 156]
  Week 92 | -17.2 [-78 to 355] | 9.3 [-94 to 125]

11. Secondary Outcome: Percent Change From Baseline in Alpha (A) 1-Microglobulin
Description: The percent change in A1-microglobulin was calculated as [Week 44 or 92 A1-microglobulin minus Baseline A1-microglobulin] divided by Baseline A1-microglobulin, multiplied by 100. For the Week 44 analysis, the last available value on/before Week 44 was used in the calculation. For the Week 92 analysis, the last available value on/before Week 92 was used in the calculation.
Time Frame: Baseline and Weeks 44, 92
Population: as for outcome 10
Measure: Median (Full Range); unit: percent change
Arm/Group | Ibandronate | Zoledronate
Number analyzed (Participants) | 38 | 37
percent change
  Week 44 | 0.0 [-85 to 706] | 0.0 [-86 to 429]
  Week 92 | 0.0 [-85 to 706] | 0.0 [-86 to 591]

12. Secondary Outcome: Percent Change From Baseline in Gamma-Glutamyltransferase (GGT)
Description: The percent change in GGT was calculated as [Week 44 or 92 GGT minus Baseline GGT] divided by Baseline GGT, multiplied by 100. For the Week 44 analysis, the last available value on/before Week 44 was used in the calculation. For the Week 92 analysis, the last available value on/before Week 92 was used in the calculation.
Time Frame: Baseline and Weeks 44, 92
Population: as for outcome 10
Measure: Median (Full Range); unit: percent change
Arm/Group | Ibandronate | Zoledronate
Number analyzed (Participants) | 38 | 37
percent change
  Week 44 | -6.0 [-57 to 393] | 3.8 [-66 to 50]
  Week 92 | -2.5 [-57 to 393] | 3.8 [-66 to 61]

13. Secondary Outcome: Percentage of Participants With Elevation of Serum Creatinine (SCr) From Baseline
Description: Elevation in SCr was defined as an increase greater than (>) 0.5 milligrams per deciliter (mg/dL) for participants with Baseline SCr less than (<) 1.4 mg/dL, or an increase >1.0 mg/dL for participants with Baseline SCr greater than or equal to (≥) 1.4 mg/dL. For the Week 44 analysis, the last available value on/before Week 44 was used. For the Week 92 analysis, the last available value on/before Week 92 was used. The percentage of participants with elevation of SCr at Weeks 44 and 92 was reported.
Time Frame: Baseline and Weeks 44, 92
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ibandronate | Zoledronate
Number analyzed (Participants) | 41 | 40
percentage of participants
  Week 44 | 2.4 [0.1 to 12.9] | 2.5 [0.1 to 13.2]
  Week 92 | 7.3 [1.5 to 19.9] | 2.5 [0.1 to 13.2]

14. Secondary Outcome: Percent Change From Baseline in CrCl
Description: CrCl was calculated from blood samples using the Cockcroft-Gault formula, and was also measured by urinalysis. The percent change in CrCl was calculated as [Week 44 or 92 CrCl minus Baseline CrCl] divided by Baseline CrCl, multiplied by 100. For the Week 44 analysis, the last available value on/before Week 44 was used in the calculation. For the Week 92 analysis, the last available value on/before Week 92 was used in the calculation.
Time Frame: Baseline and Weeks 44, 92
Population: ITT Population. The "Number of Participants Analyzed" reflects the total number of participants who provided evaluable data for the endpoint. The number of participants who provided data within the specified timeframe for each analysis (n) is shown in the table.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ibandronate | Zoledronate
Number analyzed (Participants) | 41 | 40
percent change
  Week 44, Calculated/Blood (n=41,40) | -0.5 (28.5) | -0.4 (21.7)
  Week 44, Measured/Urinalysis (n=37,37) | 6.9 (53.0) | 3.9 (37.3)
  Week 92, Calculated/Blood (n=41,40) | -0.7 (31.9) | -4.3 (20.3)
  Week 92, Measured/Urinalysis (n=37,37) | 3.1 (45.6) | 2.0 (39.1)

ADVERSE EVENTS:
Time Frame: From Baseline to end of study (up to Week 96)
Description: Safety Population: All participants who received at least one dose of study medication and completed at least one follow-up assessment visit.
Arm/Group | Ibandronate | Zoledronate
Serious Adverse Events (participants affected / at risk) | 27/46 | 18/43
Other Adverse Events (participants affected / at risk) | 43/46 | 34/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate (N=46) | Zoledronate (N=43)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Abscess oral (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Implant site infection (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 3 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 1
Septic shock (Infections and infestations) | 2 | 1
Urosepsis (Infections and infestations) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 3 | 1
Creatinine renal clearance decreased (Investigations) | 2 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate (N=46) | Zoledronate (N=43)
Anaemia (Blood and lymphatic system disorders) | 11 | 11
Leukopenia (Blood and lymphatic system disorders) | 10 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 3
Vertigo (Ear and labyrinth disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 10 | 8
Nausea (Gastrointestinal disorders) | 6 | 9
Constipation (Gastrointestinal disorders) | 4 | 4
Vomiting (Gastrointestinal disorders) | 4 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 3
Oedema peripheral (General disorders) | 7 | 10
Fatigue (General disorders) | 7 | 7
Pyrexia (General disorders) | 6 | 7
Pain (General disorders) | 4 | 4
Chills (General disorders) | 1 | 3
Chest pain (General disorders) | 0 | 3
General physical health deterioration (General disorders) | 3 | 0
Nasopharyngitis (Infections and infestations) | 19 | 10
Bronchitis (Infections and infestations) | 8 | 3
Candidiasis (Infections and infestations) | 4 | 5
Herpes zoster (Infections and infestations) | 2 | 7
Influenza (Infections and infestations) | 4 | 2
Pneumonia (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Pathological fracture (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Polyneuropathy (Nervous system disorders) | 3 | 6
Paraesthesia (Nervous system disorders) | 5 | 3
Headache (Nervous system disorders) | 5 | 2
Dizziness (Nervous system disorders) | 3 | 3
Dysgeusia (Nervous system disorders) | 3 | 0
Sleep disorder (Psychiatric disorders) | 2 | 3
Insomnia (Psychiatric disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 5
Erythema (Skin and subcutaneous tissue disorders) | 0 | 4

LIMITATIONS AND CAVEATS:
The Study was terminated as a result of slow recruitment. At the time of the decision to halt recruitment, the treatment duration was shortened to 40 weeks (instead of 92 weeks) for those participants who had not yet reached Week 48.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.